CLINICAL TRIAL: NCT05795166
Title: A Multicentre, Observational Study to Understand the Distribution of Obesity Classes and Obesity Related Comorbidities (ORCs) in People With Obesity Within a Real World Population in Czech Republic, Hungary and Poland
Brief Title: A Study to Understand the Distribution of Obesity Classes and Obesity Related Diseases in People With Obesity Across Countries in Czech Republic, Hungary and Poland
Acronym: ExplorEUEast
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-7530; U1111-1277-8275 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People with obesity: Patients with obesity coming into the clinic as part of routine visit to their treating physician/general practitioner
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
The study is intended to understand the distribution of different obesity classes and obesity related diseases (diseases that present along with obesity) in patients with body mass index (BMI) ≥ 30 kg/m^2.

Participants will be asked to give information about their health. They will continue their normal way of life and will not get any medication or additional medical test other than those prescribed to you by their doctor. Participation in the study will last for about 1 day.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Male or female, age greater than or equal to 18 years at the time of inclusion/enrolment in the study.
3. BMI greater than or equal to 30 Kg/m^2 as measured at the inclusion in the study

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study.
2. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation as judged by physician.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with obesity coming into the clinic as part of routine visit to their treating physician/general practitioner
Sampling Method: Non-Probability Sample
Enrollment: 1241 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with at least one obesity related comorbidity of interest for obesity classes I, II and III pooled across all countries | At the time of enrolment (Day 1)
  % patients with obesity

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com